CLINICAL TRIAL: NCT00662038
Title: An Open-Label Extension Study of the Long Term Safety of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Open-Label Study of the Long Term Safety of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Acronym: PIPF-012
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIPF-012; GA29960 (Other: Genentech)
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: idiopathic; pulmonary; fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): pirfenidone
  Interventions: Drug: pirfenidone

INTERVENTIONS:
Drug: pirfenidone — Pirfenidone, 2403 mg/d, administered as 801-mg doses, three times daily.

SUMMARY:
This is an open-label, multi-center, extension study for patients with IPF who complete a qualifying InterMune clinical trial of pirfenidone. The purpose of this study is to obtain additional safety data for pirfenidone 2403 mg/day in patients with IPF who complete a qualifying InterMune clinical trial of pirfenidone.

DETAILED DESCRIPTION:
This is an open-label, multi-center, extension study for patients with IPF who complete a qualifying InterMune clinical trial of pirfenidone. Eligible patients must complete the final visit for their qualifying study, have not permanently discontinued study drug in their qualifying study, and meet all of the eligibility criteria noted in this protocol.

Since data from the qualifying study may remain blinded during patient enrollment in PIPF-012, all patients will be treated as if they were taking placebo in their qualifying study. At the start of PIPF-012 participation, each patient will escalate the dose of pirfenidone.

The duration of treatment for each patient will vary and will continue until pirfenidone is commercially or otherwise available in his/her geographic region or the study is terminated by the sponsor for reasons outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Completes the qualifying clinical study final visit
* In the opinion of the principal investigator (PI), has been generally compliant with study requirements during the qualifying study, or must be considered eligible to enroll in PIPF-012 by the InterMune medical monitor
* Is able to provide informed consent and comply with the requirements of the study

Exclusion Criteria:

* Is pregnant or lactating
* Has known hypersensitivity to any of the components of the study drug
* Starts participation in another interventional clinical trial between the end of participation in the qualifying InterMune clinical trial and entry into PIPF-012
* Receives concomitant and/or excluded medications as defined in the protocol
* Permanently discontinues study drug during the qualifying study for any reason before study completion

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1058 (Actual)
Dates: Start 2008-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Genentech, Inc., South San Francisco, California, United States

REFERENCES:
- [Derived] Behr J, Nathan SD, Costabel U, Albera C, Wuyts WA, Glassberg MK, Haller H Jr, Alvaro G, Gilberg F, Samara K, Lancaster L. Efficacy and Safety of Pirfenidone in Advanced Versus Non-Advanced Idiopathic Pulmonary Fibrosis: Post-Hoc Analysis of Six Clinical Studies. Adv Ther. 2023 Sep;40(9):3937-3955. doi: 10.1007/s12325-023-02565-3. Epub 2023 Jun 30. PMID 37391667
- [Derived] Maher TM, Lancaster LH, Jouneau S, Morrison L, Lederer DJ, Molina-Molina M, Bendstrup E, Kirchgaessler KU, Gilberg F, Axmann J, Petzinger U, Noble PW. Pirfenidone Treatment in Individuals with Idiopathic Pulmonary Fibrosis: Impact of Timing of Treatment Initiation. Ann Am Thorac Soc. 2019 Jul;16(7):927-930. doi: 10.1513/AnnalsATS.201810-720RL. No abstract available. PMID 30950636
- [Derived] Costabel U, Albera C, Lancaster LH, Lin CY, Hormel P, Hulter HN, Noble PW. An Open-Label Study of the Long-Term Safety of Pirfenidone in Patients with Idiopathic Pulmonary Fibrosis (RECAP). Respiration. 2017;94(5):408-415. doi: 10.1159/000479976. Epub 2017 Sep 13. PMID 28898890
- [Derived] Lancaster L, Albera C, Bradford WZ, Costabel U, du Bois RM, Fagan EA, Fishman RS, Glaspole I, Glassberg MK, King TE Jr, Lederer DJ, Lin Z, Nathan SD, Pereira CA, Swigris JJ, Valeyre D, Noble PW. Safety of pirfenidone in patients with idiopathic pulmonary fibrosis: integrated analysis of cumulative data from 5 clinical trials. BMJ Open Respir Res. 2016 Jan 12;3(1):e000105. doi: 10.1136/bmjresp-2015-000105. eCollection 2016. PMID 26835133

RESULTS

PARTICIPANT FLOW:
Groups:
- Pirfenidone: Pirfenidone, 2403 milligrams per day (mg/d), administered orally, as capsules in 801 mg doses, three times daily.
Period: Overall Study
Arm/Group | Pirfenidone
Started | 1058
Completed | 427
Not Completed | 631
Not completed — Reason not specified | 3
Not completed — Withdrawn consent | 22
Not completed — Withdrawal by Subject | 83
Not completed — Sponsor decision | 1
Not completed — Physician Decision | 19
Not completed — Lung transplantation | 44
Not completed — Lost to Follow-up | 1
Not completed — Death | 95
Not completed — Adverse Event | 358
Not completed — Continued treatment | 5

BASELINE CHARACTERISTICS:
Population: All treated participants
Arm/Group | Pirfenidone
Number analyzed (Participants) | 1058
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (7.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 268
  Male | 790

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event defined as any unfavorable, harmful, or pathologic change in a research participant administered a pharmaceutical study treatment as indicated by physical signs, symptoms, and/or clinically significant laboratory abnormalities that occurred during the treatment and the post-treatment period, regardless of suspected cause.
Time Frame: 7.5 years
Population: All participants who received any pirfenidone.
Measure: Number; unit: percentage of participants
Arm/Group | Pirfenidone
Number analyzed (Participants) | 1058
percentage of participants | 98.0

ADVERSE EVENTS:
Time Frame: 7.5 years
Description: Adverse events were recorded at every contact with the participant.
Arm/Group | Pirfenidone
Serious Adverse Events (participants affected / at risk) | 571/1058
Other Adverse Events (participants affected / at risk) | 1027/1058
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone (N=1058)
Anaemia (Blood and lymphatic system disorders) | 5
Coagulopathy (Blood and lymphatic system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 7
Acute myocardial infarction (Cardiac disorders) | 12
Acute right ventricular failure (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 6
Angina unstable (Cardiac disorders) | 4
Aortic valve stenosis (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 26
Atrial flutter (Cardiac disorders) | 3
Atrial tachycardia (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 3
Atrioventricular block second degree (Cardiac disorders) | 4
Bradycardia (Cardiac disorders) | 5
Cardiac arrest (Cardiac disorders) | 9
Cardiac failure (Cardiac disorders) | 5
Cardiac failure acute (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 12
Cardiomyopathy (Cardiac disorders) | 1
Cor pulmonale (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 20
Coronary artery dissection (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Heart valve incompetence (Cardiac disorders) | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 7
Myocardial ischaemia (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Right ventricular dysfunction (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 4
Sick sinus syndrome (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 2
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Adrenal mass (Endocrine disorders) | 1
Eye disorder (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Abdominal adhesions (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Colonic fistula (Gastrointestinal disorders) | 2
Colonic polyp (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5
Gastrointestinal necrosis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 3
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Inguinal hernia strangulated (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 3
Intra-abdominal haematoma (Gastrointestinal disorders) | 1
Jejunal perforation (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Obstruction gastric (Gastrointestinal disorders) | 1
Oesophageal perforation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 2
Peritonitis (Gastrointestinal disorders) | 1
Rectal polyp (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3
Small intestinal perforation (Gastrointestinal disorders) | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Chest pain (General disorders) | 15
Death (General disorders) | 2
Hypothermia (General disorders) | 1
Multi-organ failure (General disorders) | 3
Non-cardiac chest pain (General disorders) | 6
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Sudden death (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 3
Cholecystitis acute (Hepatobiliary disorders) | 4
Cholecystitis chronic (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Anaphylactic reaction (Immune system disorders) | 1
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1
Polyarteritis nodosa (Immune system disorders) | 1
Abdominal abscess (Infections and infestations) | 2
Abscess intestinal (Infections and infestations) | 1
Acute sinusitis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 2
Bacterial abscess central nervous system (Infections and infestations) | 1
Bartonellosis (Infections and infestations) | 1
Bronchiectasis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 32
Bronchitis viral (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Bursitis infective (Infections and infestations) | 1
Campylobacter intestinal infection (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Cellulitis staphylococcal (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 4
Endocarditis (Infections and infestations) | 1
Endocarditis enterococcal (Infections and infestations) | 1
Enterococcal bacteraemia (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Fungal oesophagitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 1
Herpes zoster oticus (Infections and infestations) | 1
Influenza (Infections and infestations) | 7
Liver abscess (Infections and infestations) | 2
Lobar pneumonia (Infections and infestations) | 4
Lower respiratory tract infection (Infections and infestations) | 4
Lower respiratory tract infection bacterial (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Lung infection pseudomonal (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 90
Pneumonia bacterial (Infections and infestations) | 2
Pneumonia herpes viral (Infections and infestations) | 1
Pneumonia influenzal (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 4
Pneumonia streptococcal (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Postoperative abscess (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 3
Sepsis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 8
Viral infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Device lead damage (Injury, poisoning and procedural complications) | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Failure of implant (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 5
Femur fracture (Injury, poisoning and procedural complications) | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 4
Humerus fracture (Injury, poisoning and procedural complications) | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 2
Post procedural complication (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Renal haematoma (Injury, poisoning and procedural complications) | 1
Renal injury (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3
Spinal cord injury (Injury, poisoning and procedural complications) | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1
Struck by lightning (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Tendon rupture (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 2
Mycobacteria blood test positive (Investigations) | 1
Panel-reactive antibody increased (Investigations) | 1
Pulmonary arterial pressure increased (Investigations) | 1
Troponin increased (Investigations) | 1
Tumour marker increased (Investigations) | 1
Cachexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 6
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4
Hypovolaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anoxic encephalopathy (Nervous system disorders) | 1
Brain stem infarction (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 2
Central nervous system lesion (Nervous system disorders) | 1
Cerebral haematoma (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cerebral thrombosis (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 14
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 3
Demyelinating polyneuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Mononeuropathy multiplex (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Paraparesis (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 20
Syncope vasovagal (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Thalamic infarction (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 8
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Major depression (Psychiatric disorders) | 2
Psychotic disorder (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 3
Nephrolithiasis (Renal and urinary disorders) | 6
Renal cyst (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 4
Renal failure acute (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Endometriosis (Reproductive system and breast disorders) | 1
Endosalpingiosis (Reproductive system and breast disorders) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 30
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 17
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 230
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8
Pneumothorax spontaneous tension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 19
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 11
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 29
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Air embolism (Vascular disorders) | 1
Aortic aneurysm (Vascular disorders) | 4
Aortic stenosis (Vascular disorders) | 2
Arterial occlusive disease (Vascular disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 7
Embolism venous (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 7
Orthostatic hypotension (Vascular disorders) | 3
Peripheral vascular disorder (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Vasculitis necrotising (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone (N=1058)
Cataract (Eye disorders) | 53
Abdominal pain (Gastrointestinal disorders) | 60
Abdominal pain upper (Gastrointestinal disorders) | 66
Constipation (Gastrointestinal disorders) | 118
Diarrhoea (Gastrointestinal disorders) | 242
Dyspepsia (Gastrointestinal disorders) | 126
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 102
Nausea (Gastrointestinal disorders) | 305
Stomach discomfort (Gastrointestinal disorders) | 53
Vomiting (Gastrointestinal disorders) | 122
Asthenia (General disorders) | 65
Chest pain (General disorders) | 64
Fatigue (General disorders) | 210
Oedema peripheral (General disorders) | 128
Pyrexia (General disorders) | 60
Bronchitis (Infections and infestations) | 254
Influenza (Infections and infestations) | 75
Lower respiratory tract infection (Infections and infestations) | 67
Nasopharyngitis (Infections and infestations) | 202
Pneumonia (Infections and infestations) | 88
Respiratory tract infection (Infections and infestations) | 57
Sinusitis (Infections and infestations) | 130
Upper respiratory tract infection (Infections and infestations) | 295
Urinary tract infection (Infections and infestations) | 103
Weight decreased (Investigations) | 153
Anorexia (Metabolism and nutrition disorders) | 120
Decreased appetite (Metabolism and nutrition disorders) | 95
Arthralgia (Musculoskeletal and connective tissue disorders) | 89
Back pain (Musculoskeletal and connective tissue disorders) | 146
Pain in extremity (Musculoskeletal and connective tissue disorders) | 67
Dizziness (Nervous system disorders) | 176
Headache (Nervous system disorders) | 157
Syncope (Nervous system disorders) | 55
Anxiety (Psychiatric disorders) | 84
Depression (Psychiatric disorders) | 82
Insomnia (Psychiatric disorders) | 111
Cough (Respiratory, thoracic and mediastinal disorders) | 330
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 325
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 68
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 64
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 73
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 221
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 56
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 71
Productive cough (Respiratory, thoracic and mediastinal disorders) | 62
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 123
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 74
Pruritus (Skin and subcutaneous tissue disorders) | 71
Rash (Skin and subcutaneous tissue disorders) | 156
Hypertension (Vascular disorders) | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.